CLINICAL TRIAL: NCT01987596
Title: Prospective and Randomized Study of Fixed Versus Flexible Prophylactic Administration of Granulocyte Colony-Stimulating Factor (G-CSF) in Children With Cancer
Brief Title: Study of Fixed vs. Flexible Filgrastim to Accelerate Bone Marrow Recovery After Chemotherapy in Children With Cancer
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Barbara Ann Karmanos Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Children's Hospital of Michigan (Other)
Responsible Party: Principal Investigator, Maxim Yankelevich, Principal Investigator, Barbara Ann Karmanos Cancer Institute
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: 2013-062; NCI-2013-02001 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2013-062 (Other: Barbara Ann Karmanos Cancer Institute); P30CA022453 (NIH)
Record Dates: First submitted 2013-11-12; First posted 2013-11-19 (Estimated); Results first posted 2020-10-29 (Actual); Last update posted 2020-10-29 (Actual); Status verified 2020-10

CONDITIONS: Childhood Choroid Plexus Tumor; Childhood Medulloblastoma; Childhood Pineoblastoma; Childhood Soft Tissue Sarcoma; Childhood Supratentorial Primitive Neuroectodermal Tumor; Neuroblastoma; Osteosarcoma; Retinoblastoma; Wilms Tumor and Other Childhood Kidney Tumors; Recurrent/Refractory Childhood Hodgkin Lymphoma; Unspecified Childhood Solid Tumor, Protocol Specific
MeSH Terms: conditions — Choroid Plexus Neoplasms; Medulloblastoma; Neuroblastoma; Osteosarcoma; Retinoblastoma; Wilms Tumor; Recurrence | interventions — Filgrastim; Granulocyte Colony-Stimulating Factor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (fixed filgrastim) (Experimental): Patients receive filgrastim SC QD started at 24 hours after completion of chemotherapy and stopped when ANC reaches at least 1,000/uL post nadir.
  Interventions: Biological: filgrastim
- Arm II (flexible filgrastim) (Experimental): Patients receive filgrastim SC QD started on the first day after chemotherapy when ANC falls below 1,000/uL and stopped when ANC reaches at least 1,000/uL post nadir.
  Interventions: Biological: filgrastim

INTERVENTIONS:
Biological: filgrastim — Given SC once daily starting on day 1 after chemotherapy in Arm I (fixed) and on any day when ANC drops below 1000/mcl in Arm II (flexible)
  Other Names: G-CSF; Neupogen

SUMMARY:
This randomized phase III trial studies flexible administration of filgrastim after combination chemotherapy to see how well it works compared to fixed administration of filgrastim in decreasing side effects of chemotherapy in younger patients with cancer. Cancer chemotherapy frequently results in neutropenia (low blood counts) when patients are susceptible to severe infections. A medicine called G-CSF (filgrastim) stimulates bone marrow and daily filgrastim shots are commonly used to shorten neutropenic periods and decrease infections after chemotherapy. Since filgrastim is customarily used on a fixed schedule starting early after chemotherapy and there are data that early doses may not be needed, this study tests new flexible schedule of filgrastim to optimize its use by reducing the number of painful shots, cost of treatment, and filgrastim side effects in children with cancer receiving chemotherapy.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To compare the effect of flexible vs. fixed administration of G-CSF (filgrastim) on the parameters of hematological recovery including duration of absolute neutrophil count (ANC) < 500/uL; time to ANC recovery >= 1,000/uL and time to platelet recovery >= 75,000/uL in children receiving myelotoxic chemotherapy.

SECONDARY OBJECTIVES:

I. To compare the effect of flexible vs. fixed administration of G-CSF on the incidence of febrile neutropenia and number of hospital days on antibiotics following myelotoxic chemotherapy.

II. To evaluate the number of days of platelet transfusion events after chemotherapy cycles with flexible vs. fixed administration of G-CSF.

III. To evaluate on the incidence and duration of G-CSF-related side effects including extremities/back pain and headaches after chemotherapy courses followed by flexible vs. fixed administration of G-CSF.

IV. To evaluate the peripheral blood progenitor responses and subsets of progenitor cells (cluster of differentiation [CD]34/41/61/117/10/19/11b/33) to chemotherapy followed by flexible vs. fixed administration of G-CSF.

OUTLINE:

CHEMOTHERAPY: Depending on their diagnosis patients are assigned to 1 of 3 chemotherapy regimens.

ICE: Patients receive etoposide intravenously (IV) over 1 hour on days 1-3, ifosfamide IV over 3 hours on days 1-3, and carboplatin IV over 1 hour on day 4. Patients with recurrent Hodgkin lymphoma receive etoposide and ifosfamide on days 1-3 and carboplatin on day 3.

ICT: Patients receive topotecan hydrochloride IV over 30 minutes on days 1-3, and ifosfamide and carboplatin as in ICE.

OPEC: Patients receive vincristine sulfate on days 1, 8, and 15; etoposide IV over 1 hour on days 1-3; cyclophosphamide IV over 1 hour on days 1-2; and cisplatin IV over 6 hours on day 4.

For all chemotherapy regimens, treatment repeats every 21 days for 2 courses. Patients are then randomized to 1 of 2 treatment arms.

ARM I (fixed filgrastim): Patients receive filgrastim subcutaneously (SC) once daily (QD) started at 24 hours after completion of chemotherapy and stopped when ANC reaches at least 1,000/uL post nadir.

ARM II (flexible filgrastim): Patients receive filgrastim SC QD started on the first day after chemotherapy when ANC falls below 1,000/uL and stopped when ANC reaches at least 1,000/uL post nadir.

After completion of the first filgrastim treatment, patients cross-over to the other filgrastim arm and repeat the same course of chemotherapy as before. After completion of the second filgrastim treatment, chemotherapy treatment may continue for up to 5 (OPEC) or 6 (ICE, ICT) courses in the absence of disease progression or unacceptable toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have or have had at initial diagnosis, histologic proof of their malignancy; young children with primary embryonal brain tumor treated according to Head Start protocol are eligible; subjects with bone marrow involvement are NOT eligible for study
* Patients will receive repeated cycles of identical chemotherapy that will likely result in grades III-IV hematological toxicity; patients will be treated outside of Children's Oncology Group (COG) protocols with specific requirements for schedule of G-CSF administration; the following categories of patients treated at Children's Hospital of Michigan are eligible for this study:

  * Patients with brain tumors treated according to Head Start II protocol with vincristine, etoposide, cyclophosphamide, and cisplatin (OPEC) chemotherapy;
  * Patients with recurrent Hodgkin lymphoma treated with ICE (ifosfamide, carboplatin, etoposide) chemotherapy;
  * Patients with recurrent solid tumors including sarcomas, Wilms' tumor, neuroblastomas, or brain tumors treated with high dose ICE or ICT (ifosfamide, carboplatin, topotecan) chemotherapy
  * Patients with UH Wilms' tumor treated with CE (cyclophosphamide, etoposide); patients with neuroblastoma treated with CE (carboplatin, etoposide);
  * Patients with soft tissue sarcomas treated with IA (ifosfamide, doxorubicin);
  * Patients with osteosarcoma treated with high dose ifosfamide
* Subjects must have fully recovered from the toxic effects of any prior therapy; at least 3 weeks should have elapsed since the last dose of chemotherapy (6 weeks in the case of nitrosourea containing therapy); subjects must have recovered from previous colony-stimulating factor therapy and have been off colony-stimulating factors (G-CSF, granulocyte macrophage colony-stimulating factor [GM-CSF], interleukin [IL]-11) for more than 10 days and off erythropoietin for 30 days
* ANC > 1000/uL
* Platelet count > 100,000/uL
* Creatinine clearance or glomerular filtration rate (GFR) which is greater than or equal to 70 ml/min/1.73 m^2
* Bilirubin less than 1.5 x normal limit (NL)
* Serum glutamic oxaloacetic transaminase (SGOT) or serum glutamate pyruvate transaminase (SGPT) less than 2.5 x NL for age
* Subjects should have a normal ejection fraction (per institutional limits), no evidence of cardiac arrhythmias requiring therapy, and a fractional shortening of > 28%
* All subjects must have a life expectancy of 12 weeks or more
* Diagnostic categories

  * Sarcoma (soft tissue and bone)
  * Kidney tumors
  * Brain tumors
  * Other solid tumors (gonadal and germ cell tumors, retinoblastoma, neuroblastoma, and miscellaneous tumors)
  * Hodgkin lymphoma
* Performance status must be > 60 from Lansky (age 1 to 16) or Karnofsky (age > 16)

Exclusion Criteria:

* Subjects with any of the following will NOT be eligible for study:

  * Bone marrow involvement
  * Active myelogenous leukemia, or history of myelogenous leukemia
  * Pregnancy

Ages: 1 Year to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 23 (Actual)
Dates: Start 2013-08; Primary Completion 2018-06 (Actual); Study Completion 2018-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Maxim Yankelevich, Principal Investigator — Barbara Ann Karmanos Cancer Institute
Locations (1):
- Barbara Ann Karmanos Cancer Institute, Detroit, Michigan, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm I (Fixed Flexible Filgrastim Schedule): Period 1 Fixed: Patients receive filgrastim SC QD once daily started at 24 hours after completion of chemotherapy and stopped when ANC reaches at least 1,000/uL post nadir.
  Period 2 Flexible: Patients receive filgrastim:SC once starting on day 1 after chemotherapy in Arm I (fixed) and on any day when ANC drops below 1000/mcl in Arm II (flexible)
- Arm II (Flexible Fixed Filgrastim Schedule): Period 1 Flexible: Patients receive filgrastim SC QD started on the first day after chemotherapy and on any day when ANC falls below 1,000/uL and stopped when ANC reaches at least 1,000/uL post nadir.
  Period 2 Fixed: Patients receive filgrastim: given SC once daily starting on day 1 after chemotherapy in and daily thereafter until ANC reaches at least 1,000/uL post nadir.
Period: Overall Study
Arm/Group | Arm I (Fixed Flexible Filgrastim Schedule) | Arm II (Flexible Fixed Filgrastim Schedule)
Started | 12 | 11
Completed | 11 | 10
Not Completed | 1 | 1
Not completed — Physician Decision | 1 | 0
Not completed — Progressive Disease; missing all period | 0 | 1

BASELINE CHARACTERISTICS:
Population: All participants who completed period 2
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I (Fixed Flexible Filgrastim Schedule) | Arm II (Flexible Fixed Filgrastim Schedule) | Total
Number analyzed (Participants) | 11 | 10 | 21
Age, Continuous [Median (Full Range); unit: years] | 16 [6 to 22] | 11 [5 to 22] | 14 [5 to 22]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 5 | 7
  Male | 9 | 5 | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 10 | 10 | 20
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 4 | 8
  White | 4 | 5 | 9
  More than one race | 3 | 0 | 3
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 11 | 10 | 21

OUTCOME MEASURES:

1. Primary Outcome: Days to ANC Greater Than or Equal to 1,000/uL From the Start of Chemotherapy
Description: Time in days until absolute neutrophil count (ANC) recovery to greater than or equal to 1,000/uL from the start of chemotherapy
Time Frame: From the start of the course until the first date the ANC reaches >= 1,000/uL post nadir, assessed up to 1 year
Measure: Mean (95% Confidence Interval); unit: days
Groups:
- Fixed: Mean of time to ANC1000 during period participants were on fixed regimen
- Flexible: Mean of time to ANC1000 during period participants were on flexible regimen
Arm/Group | Fixed | Flexible
Number analyzed (Participants) | 21 | 21
days | 16.0 [15.0 to 17.1] | 16.7 [15.7 to 17.7]

2. Secondary Outcome: Incidence of Febrile Neutropenia
Description: occurrence of febrile neutropenia
Time Frame: Up to 1 year
Population: Each patient server as his/her own control
Measure: Count of Participants; unit: Participants
Groups:
- Fixed: Incidence duriing time patient was on fixed schedule
- Flexible: Incidence duriing time patient was on flexible schedule
Arm/Group | Fixed | Flexible
Number analyzed (Participants) | 21 | 21
Participants
  Yes | 5 | 6
  No | 16 | 15
Statistical Analysis 1: Comparison: Fixed vs Flexible; Test type: Superiority; p = 1.00, McNemar

3. Secondary Outcome: Cumulative GCSF Dose
Description: Cumulative GCSF dose - number of GCSF injections until ANC recovery greater than or equal to 1,000/uL from the start of chemotherapy
Time Frame: up until engraftment
Population: Patients who had data for period 2
Measure: Mean (95% Confidence Interval); unit: Doses
Groups:
- Fixed Filgrastim: Patients receive filgrastim daily SC QD started at 24 hours after completion of chemotherapy and stopped when ANC reaches at least 1,000/uL post nadir.
- Flexible Filgrastim: Patients receive filgrastim SC QD started on the first day after chemotherapy and on any day ANC falls below 1,000/uL and stopped when ANC reaches at least 1,000/uL post nadir.
Arm/Group | Fixed Filgrastim | Flexible Filgrastim
Number analyzed (Participants) | 19 | 19
Doses | 10.5 [9.6 to 11.2] | 6.7 [5.5 to 7.9]
Statistical Analysis 1: Comparison: Fixed Filgrastim vs Flexible Filgrastim; two-period crossover design analysis; Test type: Superiority; p < 0.0001, ANOVA

4. Secondary Outcome: Days to First G-CSF Dose
Description: Time (in days) to first G-CSF dose
Time Frame: time to ANC 1000
Population: All participants with period 2 data
Measure: Mean (95% Confidence Interval); unit: days
Groups:
- Arm I (Fixed Filgrastim): Patients receive filgrastim SC QD started at 24 hours after completion of chemotherapy and continued daily until ANC reaches at least 1,000/uL post nadir.
Arm/Group | Arm I (Fixed Filgrastim) | Arm II (Flexible Filgrastim)
Number analyzed (Participants) | 19 | 19
days | 5.1 [4.5 to 5.7] | 9.5 [8.4 to 10.5]
Statistical Analysis 1: Comparison: Arm I (Fixed Filgrastim) vs Arm II (Flexible Filgrastim); 2 treatment, 2 periiod cross-over analysis; Test type: Superiority; p < 0.0001, ANOVA

ADVERSE EVENTS:
Time Frame: 6 months
Description: Nothing to mention
Arm/Group | Arm I (Fixed Filgrastim) | Arm II (Flexible Filgrastim)
All-Cause Mortality (participants affected / at risk) | 0/21 | 0/21
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/21
Other Adverse Events (participants affected / at risk) | 4/21 | 1/21
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (Fixed Filgrastim) (N=21) | Arm II (Flexible Filgrastim) (N=21)
Pain (Nervous system disorders) | 4 (6) | 1 (2) — GCSF related pain (headaches, back or extremities pain)
Pain (Nervous system disorders) | 4 (6) | 1 (2) — GCSF related pain including headaches, back and extremities pain

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2013-11-14): https://cdn.clinicaltrials.gov/large-docs/96/NCT01987596/Prot_SAP_000.pdf